CLINICAL TRIAL: NCT07047261
Title: Efficacy of a Xanthan-based Chlorhexidine Gel in the Treatment of Peri-implant Mucositis: a Randomized Split-mouth Clinical Trial
Brief Title: Efficacy of a Xanthan-based Chlorhexidine Gel in the Treatment of Peri-implant Mucositis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jacopo Lanzetti, Dental Hygienist Registered (RDH), University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00453/2024
Record Dates: First submitted 2025-06-17; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Peri-implant Mucositis
Keywords: Peri-implant mucositis; adjunctive treatment; professional mechanical plaque removal; Xanthan-chlorhexidine based gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional mechanical plaque removal with xanthan-chlorhexidine based gel (Experimental): At baseline, after recording clinical parameters, patients received oral hygiene instruction and underwent periodontal debridement alternating ultrasonic with manual instruments, followed by the use of air-abrasive devices with 25-micron glycine powder and a supragingival tip Subsequently, the clinician cleaned and dried the site using compressed air and applied the XanCHX gel on the implant sites assigned to the test group, positioning the blunt needle at the bottom of the pocket and gently extruding the product while moving it out of the site. Finally, the patient was instructed not to drink or rinse for the following hour. At each time-step, clinical assessments were recorded after the reinforcement in oral hygiene instruction and professional implant hygiene using rubber cup and polishing paste.
  Interventions: Procedure: Adjunctive use of Xanthan-Chlorexidine based gel
- Professional mechanical plaque removal alone (No Intervention): At baseline, after recording clinical parameters, patients received oral hygiene instruction and underwent periodontal debridement alternating ultrasonic with manual instruments, followed by the use of air-abrasive devices with 25-micron glycine powder and a supragingival tip. At each time-step, clinical assessments were recorded after the reinforcement in oral hygiene instruction and professional implant hygiene using rubber cup and polishing paste.

INTERVENTIONS:
Procedure: Adjunctive use of Xanthan-Chlorexidine based gel — The chlorhexidine and xanthan-based gel contains 0.5% chlorhexidine digluconate, 1% chlorhexidine dihydrochloride, and 0.5% xanthan gel. Xanthan is a polymer that creates a three-dimensional, pseudo-plastic network with water, forming a stable gel that allows a slow and prolonged release of chlorhexidine, allowing effectiveness for about 30 days. Chlorhexidine digluconate is released immediately upon application, whereas Chlorhexidine dihydrochloride is gradually delivered the following days, providing bacteriostatic and bactericidal effects for up to two weeks, helping the prevention of recolonization of treated site.
  The clinician cleaned and dried the implant site using compressed air and applied the XanCHX gel on the implant sites assigned to the test group, positioning the blunt needle at the bottom of the pocket and gently extruding the product while moving it out of the site. Finally, the patient was instructed not to drink or rinse for the following hour.
  Arms: Professional mechanical plaque removal with xanthan-chlorhexidine based gel

SUMMARY:
The peri-implant mucositis is an inflammatory and reversible lesion that surrounds the peri-implant mucosa without loss of supporting bone, clinically characterized by bleeding on gentle probing. It has been estimated that it affects approximately 21% to 88% of individuals and 9% to 51% of implant sites, with prevalences of 47% and 29%, respectively.

Experimental clinical researches show that peri-implant mucositis can be reversed if proper biofilm management is maintained. Prevention and regression of inflammation around the implant can be achieved through proper oral hygiene and an effective supportive care protocol, which may include regular clinical check-ups, radiographic assessments, oral hygiene instructions and professional mechanical plaque removal (PMPR).

Therefore, adjunctive measures such as self-administration of oral rinse antiseptics (i.e. chlorhexidine) may be considered. For examples, the use of a chlorhexidine-based gel in combination with xanthan (XanCHX), in addition to PMPR has demonstrated clinical improvements in the treatment of periodontitis.

The aim of the present study was to investigate the potential benefits of XanCHX gel in adjunction to PMPR in patients affected by peri-implant mucositis, promoting a complete healing of the affected tissues.

ELIGIBILITY:
Inclusion Criteria:

* presence of two or more peri-implant mucositis sites (e.g. presence of bleeding and/or suppuration on probing with no bone loss evident on radiographs);
* implant-supported fixed restorations inserted at least 6 months before patient enrollment

Exclusion Criteria:

* radiation therapy in the head and neck therapy or long-term corticosteroid treatments;
* use of systemic antibiotics for more than 6 months;
* diagnosis of not plaque-associated inflammatory diseases (e.g., Oral Lichen Planus);
* pregnant or breastfeeding mother;
* untreated peri-implantitis;
* oral rehabilitation with full-arch prostheses;
* allergy to chlorhexidine and/or other components contained in the gel.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding on Probing | From baseline until the end of the study (6 months)
  Presence or absence of gingival bleeding within 30 seconds after probing

SECONDARY OUTCOMES:
Probing pocket depth | From the baseline until the end of the study (6 months)
  Measure from the peri-implant mucosal margin to the base of the sulcus, applying a force of 0.2 N (20g)
Plaque index | From baseline until the end of the study (6 months)
  Presence or absence of plaque on implant surfaces
Gingival recession | From the baseline until the end of the study (6 months)
  Measure from prosthetic crown to the peri-implant mucosal margin in millimeters
Keratinized gingiva | From the baseline until the end of the study (6 months)
  Measure from the peri-implant mucosal margin to oral mucosal margin in millimeters
Clinical attachment level | From the baseline until the end of the study (6 months)
  Measure, in millimeters, of the amount of gum tissue and bone attached to the root of the tooth. Specifically, it is the sum of the measurement of gingival recession and the probing depth.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy, Italy